CLINICAL TRIAL: NCT07182409
Title: Efficacy and Safety of Monoclonal Antibody in Acute Phase of Neuromyelitis Optica Spectrum Disorder（MAAP-NMO），A Prospective, Multicenter Cohort Study
Brief Title: Efficacy and Safety of Monoclonal Antibody in Acute Phase of Neuromyelitis Optica Spectrum Disorder
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Feng Jinzhou, Associate professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: MAAP-NMO-001
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: NMOSD
Keywords: NMOSD; Intravenous methylprednisolone; Efgartigimod; Eculizumab; Plasma exchange

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples will be collected at four time points (baseline, month 1, month 3, and month 6).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- IVMP group: Methylprednisolone, intravenous infusion, 1000 mg/day for 5 consecutive days.
- IVMP + Plasma Exchange (PE) group: IVMP combined with plasma exchange, 2000-3000 mL per session, once every 1-2 days, for a total of 3-5 sessions.
- IVMP + Efgartigimod group: IVMP combined with efgartigimod, intravenous infusion, 10 mg/kg once weekly for 4 weeks.
- IVMP + Eculizumab group: IVMP combined with eculizumab, intravenous infusion of 900 mg once weekly for 4 weeks.

SUMMARY:
This study aims to evaluate the efficacy and safety of different monoclonal antibody in the acute phase of neuromyelitis optica spectrum disorder (MAAP-NMO). It will also examine immune-related biomarkers and their relationship with treatment response to provide evidence for optimizing acute-phase therapeutic strategies.

DETAILED DESCRIPTION:
Neuromyelitis optica spectrum disorder (NMOSD) is an inflammatory demyelinating disease of the central nervous system characterized primarily by humoral immune dysfunction. The acute phase is highly disabling; therefore, improving the effectiveness of acute-phase interventions represents a critical challenge in the clinical management of NMOSD. Conventional acute treatments such as intravenous methylprednisolone (IVMP), plasma exchange (PE), and intravenous immunoglobulin (IVIg) provide only limited rates of remission. The advent of novel biologics has expanded therapeutic options for NMOSD, but consensus regarding the optimal treatment approach during the acute phase has not yet been established.

This project is a multicenter, prospective, real-world observational study. A total of 35-45 patients with acute-phase NMOSD from 12 centers across China will be enrolled and followed systematically for at least 6 months according to a standardized protocol. The study will evaluate the real-world efficacy and safety of different monoclonal antibodies, primarily focusing on efgartigimod and eculizumab, in the treatment of acute-phase NMOSD. It will further assess their impact on symptom and neurological disability improvement, as well as their effects on immunological parameters, biomarkers, and imaging outcomes, in order to explore the optimal acute-phase immunotherapy strategy in NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Age at onset ≥18 years, any gender.
2. Patients meeting the 2015 International Panel for NMO Diagnosis (IPND) criteria for NMOSD and currently in the acute phase, defined as new or significantly worsened neurological deficits lasting >24 hours, with onset within <14 days, excluding pseudo-relapses caused by fever, infection, or metabolic disturbances. The acute relapse must meet at least one of the following clinical phenotypes: a) Optic neuritis (ON): EDSS visual function score ≥3; b) Transverse myelitis (TM): EDSS pyramidal function score ≥2. NMOSD-related syndromes (e.g., area postrema syndrome, acute brainstem syndrome, acute diencephalic syndrome, cerebral syndrome) may be present as concomitant features but cannot be the sole or primary manifestation.
3. Serum AQP4-IgG positive by cell-based assay (CBA) with a titer ≥1:32, and negative for MOG-IgG (CBA or LCBA) and GFAP-IgG.
4. Expanded Disability Status Scale (EDSS) score at enrollment ≥3 and ≤8 points.
5. Planned to receive or currently receiving intravenous methylprednisolone (IVMP) treatment, and not on or only using conventional immunosuppressive maintenance therapy.
6. Able to comply with standardized follow-up, with an expected minimum follow-up of 12 months during the study period.
7. Signed informed consent by the patient or legal guardian (if applicable).

Exclusion Criteria:

1. Participation in a randomized clinical trial with blinded treatment allocation.
2. Received treatment with monoclonal antibody (including rituximab, satralizumab, inebilizumab, eculizumab, efgartigimod, etc.) within 3 months prior to screening.
3. Received treatment with IVIg, plasma exchange (PE), IVMP, or oral corticosteroids >30 mg/day within 1 month prior to screening.
4. Incomplete or unavailable follow-up data, expected inability to complete follow-up, or poor compliance.
5. Patients who have independently discontinued immunotherapy or demonstrate poor adherence.
6. Presence of severe underlying diseases or other conditions that may affect the safety of immunotherapy or the interpretation of study results, including but not limited to: a) Chronic or active infections requiring long-term systemic treatment (e.g., progressive multifocal leukoencephalopathy, chronic renal infection, chronic respiratory infection with bronchiectasis, active tuberculosis, active hepatitis C, etc.); b) Positive hepatitis B serology (except in individuals with prior vaccination); c) History or suspicion of tuberculosis; d) Positive HIV serology; e) History or current clinically significant adverse reactions (including severe allergic reactions) related to corticosteroids, FcRn antagonists, or complement inhibitors.
7. Pregnant or breastfeeding women, or women planning pregnancy in the near future (contraception required during treatment).
8. Any other condition deemed by the investigators to make participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NMOSD patients with acute attacks
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score | 1 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline to 1 months after treatment (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score | 3 and 6 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline at 3 and 6 months (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Percentage of Participants with Improvement | 1, 3 and 6 months
  Improvement is defined as:
  1. ≥1.0-point decrease from baseline if baseline EDSS ≤5.5;
  2. ≥0.5-point decrease from baseline if baseline EDSS >5.5.
Change in Low-Contrast Visual Acuity (LCVA) | 1, 3 and 6 months
  Low-Contrast Visual Acuity (LCVA), using a standardized low-contrast ETDRS visual acuity chart, the number of letters that the patient can identify at a sitting position and a distance of 4 meters / 1 meter is measured to reflect the recovery of visual function.
Percentage of Participants without relapse | 1, 3 and 6 months
  Relapse is defined as new neurological symptoms or significant worsening of existing symptoms lasting ≥24 hours during the follow-up period, excluding causes such as infection or fever, and confirmed by imaging or clinical evaluation.
MRI changes after immunotherapy | 1 and 6 months
  MRI changes including improvement of acute-phase pre-existing T2 hyperintense lesions and enhancing lesions (volume reduction, signal attenuation, or decreased enhancement), and the number of new and/or enlarged T2 hyperintense lesions or new enhancing lesions.
Change in serum AQP4-IgG titer | 1, 3 and 6 months
  Change in serum AQP4-IgG titer before treatment and at 1, 3, and 6 months after immunotherapy, measured by cell-based assay.
Change in serum GFAP level | 1, 3, and 6 months
  Change in serum GFAP level before treatment and at 1, 3, and 6 months after immunotherapy, measured by Simoa immunoassay.
Change in serum NfL level | 1, 3, and 6 months
  Change in serum NfL level before treatment and at 1, 3, and 6 months after immunotherapy, measured by Simoa immunoassay.
Changes in serum IL-6, IL-17, TNF-α, IFN-γ, and IL-10 levels | 1, 3 and 6 months
  Changes in serum IL-6, IL-17, TNF-α, IFN-γ, and IL-10 levels before treatment and at 1, 3, and 6 months after immunotherapy, measured by multiplex bead-based immunoassay. Units: pg/mL.
Changes in T/B cell subsets | 1, 3 and 6 months
  Changes in T/B cell subsets (immune function monitoring) before treatment and at 1, 3, and 6 months after immunotherapy.
Changes in serum lactate, pyruvate, and glucose levels | 1, 3 and 6 months
  Energy metabolism will be assessed by quantifying serum lactate, pyruvate, and glucose concentrations at baseline, 1, 3, and 6 months using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Units: mmol/L.
Changes in serum lipid metabolites | 1, 3 and 6 months
  Lipid metabolism will be evaluated by measuring serum cholesterol at baseline, 1, 3 and 6 months using LC-MS/MS. Units: µmol/L.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 1, 3 and 6 months
  AEs are any unfavorable medical occurrences during the study period, regardless of causality. SAEs include events resulting in death, life-threatening conditions, permanent or significant disability or loss of function, hospitalization or prolongation of hospitalization, congenital anomaly, or birth defect. Record the time of onset, type, severity, and outcome. Drug-related adverse effects of biologics (e.g., efgartigimod, inebilizumab) will be specifically monitored, including hypogammaglobulinemia (assessed at baseline, 1, 3, and 6 months) and occurrence of meningococcal infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Feng, Ph.D, Principal Investigator — First Affiliated Hospital of Chongqing Medical University